CLINICAL TRIAL: NCT06880185
Title: Effects of Ribose Cross-Linked Thick Collagen Membranes and Connective Tissue Grafts on Peri-Implant Tissue
Brief Title: Soft Tissue Management in Peri-Implant Regions
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Ömer Alperen Kırmızıgül (Other)
Collaborators: Inonu University (Other)
Responsible Party: Sponsor-Investigator, Ömer Alperen Kırmızıgül, Assistant Prof Dr, Inonu University
Organization: Inonu University (Other)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: İNU-DHF-ŞMK-01
Record Dates: First submitted 2025-03-11; First posted 2025-03-17 (Actual); Last update posted 2025-12-09 (Actual); Status verified 2025-03

CONDITIONS: Peri-implant Mucosa Thickness; Peri-implant Mucosa Width; Peri-Implant Tissues
Keywords: Collagen membranes; Soft tissue; Peri-implant mucosa thickness; Peri-implant mucosa width; Connective tissue graft

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Control (Other): Connective Tissue Graft
  Interventions: Other: Connective Tissue Graft
- Test (Active Comparator): Ribose Cross-Linked Thick Collagen Membrane
  Interventions: Other: Ribose Cross-Linked Thick Collagen Membrane

INTERVENTIONS:
Other: Connective Tissue Graft — Implant treatment was performed in 20 patients with a single tooth deficiency and soft tissue deficiency in the horizontal direction in the edentulous site. All patients received bone-level titanium implants. Soft tissue augmentation was performed simultaneously with implant treatment. The group were divided into CTG , and 10 patients were randomly assigned to group.
  Arms: Control
Other: Ribose Cross-Linked Thick Collagen Membrane — Implant treatment was performed in 20 patients with a single tooth deficiency and soft tissue deficiency in the horizontal direction in the edentulous site. All patients received bone-level titanium implants. Soft tissue augmentation was performed simultaneously with implant treatment. The groups were divided into RCCM, and 10 patients were randomly assigned to group.
  Arms: Test

SUMMARY:
Background:This study aimed to compare the effect of ribose cross-linked thick collagen membrane (RCCM) with that of subepithelial connective tissue graft (CTG) in sites with soft tissue deficiency in the horizontal aspect around the implant.

Methods:Single implant sites were included in the study of 20 systemically healthy patients. All procedures were performed concurrently with implant placement; SCTG was administered in ten patients, and RCCM in the other ten. Before the operation, the PIMT and peri-implant mucosa width (PIMW) were measured. Visual analog scale (VAS) and Oral Health Impact profile-14 (OHIP-14) scores were recorded on post-operative days 1, 3, and 7. At 1 and 3 months measurements were repeated.

Results:In terms of PIMT, an average increase of 1.87 mm was recorded in the RCCM group and 1.99 mm in the SCTG group. The rate of increase in PIMT was statistically similar in both the groups (p>0.05). The OHIP-14 and VAS scores were similar between the groups on days 1, 3, and 7. There was a decrease at 3 months in both the groups.

Conclusion:Within the limits of this study, RCCM provided a similar increase in PIMT as SCTG. RCCM is a promising alternative to SCTG for increasing the PIMT.

Keywords: Collagen, Connective tissue, Dental implants, Oral mucosa

ELIGIBILITY:
Inclusion Criteria:

* Systemically healthy
* The edentulous space for which implant treatment is planned to be single tooth size and molar tooth site
* Those with soft tissue deficiency in the horizontal aspect in the site where implant treatment is planned
* Age between 18-60 years
* Does not have a condition that may cause a bleeding disorder
* No nausea-vomiting reflex
* Patients with good oral hygiene

Exclusion Criteria:

* Patients with systemic disorders (diabetes, hypertension, radiotherapy/ chemotherapy, etc.)
* Patients who have insufficient horizontal alveolar bone in the site where implant treatment is planned and who may lead to bone dehiscence after implant placement
* Patients with collagen allergy
* Those taking any medication that may affect wound healing
* Those with bleeding disorders
* Smokers who smoke more than 10 cigarettes a day
* Poor oral hygiene
* Those with vomiting-nausea reflex
* Allergic to anti-inflammatory drugs
* Patients with pregnancy/breastfeeding status.

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 20 (Actual)
Dates: Start 2023-12-01 (Actual); Primary Completion 2024-12-30 (Actual); Study Completion 2024-12-30 (Actual)

PRIMARY OUTCOMES:
Peri-implant Mucosa Thickness | From the beginning to the 3rd month
  Changes in peri-implant mucosal thickness at baseline, month 1 and month 3

CONTACTS AND LOCATIONS:
Locations (1):
- Inonu Unıversity Faculty of Dentistry, Malatya, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Zucchelli G, Tavelli L, Stefanini M, Barootchi S, Mazzotti C, Gori G, Wang HL. Classification of facial peri-implant soft tissue dehiscence/deficiencies at single implant sites in the esthetic zone. J Periodontol. 2019 Oct;90(10):1116-1124. doi: 10.1002/JPER.18-0616. Epub 2019 Jun 3. PMID 31087334
- [Result] Zucchelli G, Tavelli L, McGuire MK, Rasperini G, Feinberg SE, Wang HL, Giannobile WV. Autogenous soft tissue grafting for periodontal and peri-implant plastic surgical reconstruction. J Periodontol. 2020 Jan;91(1):9-16. doi: 10.1002/JPER.19-0350. Epub 2019 Oct 6. PMID 31461778
- [Result] Vallecillo C, Toledano-Osorio M, Vallecillo-Rivas M, Toledano M, Rodriguez-Archilla A, Osorio R. Collagen Matrix vs. Autogenous Connective Tissue Graft for Soft Tissue Augmentation: A Systematic Review and Meta-Analysis. Polymers (Basel). 2021 May 31;13(11):1810. doi: 10.3390/polym13111810. PMID 34072698
- [Result] Tommasato G, Del Fabbro M, Oliva N, Khijmatgar S, Grusovin MG, Sculean A, Canullo L. Autogenous graft versus collagen matrices for peri-implant soft tissue augmentation. A systematic review and network meta-analysis. Clin Oral Investig. 2024 May 5;28(5):300. doi: 10.1007/s00784-024-05684-5. PMID 38704784
- [Result] Thoma DS, Zeltner M, Hilbe M, Hammerle CH, Husler J, Jung RE. Randomized controlled clinical study evaluating effectiveness and safety of a volume-stable collagen matrix compared to autogenous connective tissue grafts for soft tissue augmentation at implant sites. J Clin Periodontol. 2016 Oct;43(10):874-85. doi: 10.1111/jcpe.12588. Epub 2016 Aug 12. PMID 27310522
- [Result] Thoma DS, Strauss FJ, Mancini L, Gasser TJW, Jung RE. Minimal invasiveness in soft tissue augmentation at dental implants: A systematic review and meta-analysis of patient-reported outcome measures. Periodontol 2000. 2023 Feb;91(1):182-198. doi: 10.1111/prd.12465. Epub 2022 Aug 11. PMID 35950734
- [Result] Thoma DS, Strauss FJ. On the discrepancy between professionally assessed and patient-reported outcome measures. J Periodontal Implant Sci. 2022 Apr;52(2):89-90. doi: 10.5051/jpis.225202edi01. No abstract available. PMID 35505571
- [Result] Thoma DS, Gasser TJW, Hammerle CHF, Strauss FJ, Jung RE. Soft tissue augmentation with a volume-stable collagen matrix or an autogenous connective tissue graft at implant sites: Five-year results of a randomized controlled trial post implant loading. J Periodontol. 2023 Feb;94(2):230-243. doi: 10.1002/JPER.22-0226. Epub 2022 Oct 28. PMID 35904229
- [Result] Tavelli L, Majzoub J, Kauffmann F, Rodriguez MV, Mancini L, Chan HL, Kripfgans OD, Giannobile WV, Wang HL, Barootchi S. Coronally advanced flap versus tunnel technique for the treatment of peri-implant soft tissue dehiscences with the connective tissue graft: A randomized, controlled clinical trial. J Clin Periodontol. 2023 Jul;50(7):980-995. doi: 10.1111/jcpe.13806. Epub 2023 Apr 4. PMID 36935199
- [Result] Tavelli L, Barootchi S, Rodriguez MV, Meneghetti PC, Mendonca G, Wang HL. Volumetric Outcomes of Peri-implant Soft Tissue Augmentation with a Xenogeneic Cross-Linked Collagen Scaffold: A Comparative Clinical Study. Int J Periodontics Restorative Dent. 2023 Jul-Aug;43(4):415-422. doi: 10.11607/prd.6058. PMID 37552200
- [Result] Tavelli L, Barootchi S, Avila-Ortiz G, Urban IA, Giannobile WV, Wang HL. Peri-implant soft tissue phenotype modification and its impact on peri-implant health: A systematic review and network meta-analysis. J Periodontol. 2021 Jan;92(1):21-44. doi: 10.1002/JPER.19-0716. Epub 2020 Aug 9. PMID 32710810
- [Result] Subramanya AP, Prabhuji MLV. Synthetic mineral collagen composite bone graft with ribose cross linked collagen membrane for lateral ridge augmentation. J Indian Soc Periodontol. 2023 May-Jun;27(3):332-335. doi: 10.4103/jisp.jisp_306_22. Epub 2023 May 1. PMID 37346848
- [Result] Stefanini M, Barootchi S, Sangiorgi M, Pispero A, Grusovin MG, Mancini L, Zucchelli G, Tavelli L. Do soft tissue augmentation techniques provide stable and favorable peri-implant conditions in the medium and long term? A systematic review. Clin Oral Implants Res. 2023 Sep;34 Suppl 26:28-42. doi: 10.1111/clr.14150. PMID 37750532
- [Result] Slade GD, Spencer AJ. Social impact of oral conditions among older adults. Aust Dent J. 1994 Dec;39(6):358-64. doi: 10.1111/j.1834-7819.1994.tb03106.x. PMID 7832683
- [Result] Scheyer ET, Sanz M, Dibart S, Greenwell H, John V, Kim DM, Langer L, Neiva R, Rasperini G. Periodontal soft tissue non-root coverage procedures: a consensus report from the AAP Regeneration Workshop. J Periodontol. 2015 Feb;86(2 Suppl):S73-6. doi: 10.1902/jop.2015.140377. PMID 25644301
- [Result] Nisanci Yilmaz MN, Koseoglu Secgin C, Ozemre MO, Inonu E, Aslan S, Bulut S. Assessment of gingival thickness in the maxillary anterior region using different techniques. Clin Oral Investig. 2022 Nov;26(11):6531-6538. doi: 10.1007/s00784-022-04602-x. Epub 2022 Jul 7. PMID 35796801
- [Result] McGuire MK, Janakievski J, Scheyer ET, Velasquez D, Gunsolley JC, Heard RH, Morelli T. Efficacy of a harvest graft substitute for recession coverage and soft tissue volume augmentation: A randomized controlled trial. J Periodontol. 2022 Mar;93(3):333-342. doi: 10.1002/JPER.21-0131. Epub 2021 Aug 16. PMID 34287902
- [Result] Levin BP, Zubery Y. Use of a Sugar Cross-Linked Collagen Membrane Offers Cell Exclusion and Ossification. Compend Contin Educ Dent. 2018 Jan;39(1):44-48. PMID 29293010
- [Result] Langer B. The regeneration of soft tissue and bone around implants with and without membranes. Compend Contin Educ Dent. 1996 Mar;17(3):268-70, 272 passim; quiz 280. PMID 9051957
- [Result] Fu JH, Yeh CY, Chan HL, Tatarakis N, Leong DJ, Wang HL. Tissue biotype and its relation to the underlying bone morphology. J Periodontol. 2010 Apr;81(4):569-74. doi: 10.1902/jop.2009.090591. PMID 20367099
- [Result] Friedmann A, Gissel K, Soudan M, Kleber BM, Pitaru S, Dietrich T. Randomized controlled trial on lateral augmentation using two collagen membranes: morphometric results on mineralized tissue compound. J Clin Periodontol. 2011 Jul;38(7):677-85. doi: 10.1111/j.1600-051X.2011.01738.x. Epub 2011 May 10. PMID 21557757
- [Result] Delgado DA, Lambert BS, Boutris N, McCulloch PC, Robbins AB, Moreno MR, Harris JD. Validation of Digital Visual Analog Scale Pain Scoring With a Traditional Paper-based Visual Analog Scale in Adults. J Am Acad Orthop Surg Glob Res Rev. 2018 Mar 23;2(3):e088. doi: 10.5435/JAAOSGlobal-D-17-00088. eCollection 2018 Mar. PMID 30211382
- [Result] De Bruyckere T, Cosyn J, Younes F, Hellyn J, Bekx J, Cleymaet R, Eghbali A. A randomized controlled study comparing guided bone regeneration with connective tissue graft to re-establish buccal convexity: One-year aesthetic and patient-reported outcomes. Clin Oral Implants Res. 2020 Jun;31(6):507-516. doi: 10.1111/clr.13587. Epub 2020 Feb 21. PMID 32011032
- [Result] Chackartchi T, Gleis R, Sculean A, Nevins M. A Novel Surgical Approach to Modify the Periodontal Phenotype for the Prevention of Mucogingival Complications Related to Orthodontic Treatment. Int J Periodontics Restorative Dent. 2021 Nov-Dec;41(6):811-817. doi: 10.11607/prd.5774. PMID 34818383
- [Result] Cairo F, Barbato L, Tonelli P, Batalocco G, Pagavino G, Nieri M. Xenogeneic collagen matrix versus connective tissue graft for buccal soft tissue augmentation at implant site. A randomized, controlled clinical trial. J Clin Periodontol. 2017 Jul;44(7):769-776. doi: 10.1111/jcpe.12750. Epub 2017 Jun 29. PMID 28548210
- [Result] Buser D, Sennerby L, De Bruyn H. Modern implant dentistry based on osseointegration: 50 years of progress, current trends and open questions. Periodontol 2000. 2017 Feb;73(1):7-21. doi: 10.1111/prd.12185. PMID 28000280
- [Result] Barootchi S, Tavelli L, Zucchelli G, Giannobile WV, Wang HL. Gingival phenotype modification therapies on natural teeth: A network meta-analysis. J Periodontol. 2020 Nov;91(11):1386-1399. doi: 10.1002/JPER.19-0715. Epub 2020 Jun 12. PMID 32392401